CLINICAL TRIAL: NCT03751527
Title: ZENFlex-Registry to Evaluate the Outcome of Bare Metal Stent-assisted Angioplasty in the Treatment of Superficial Femoral and/or Proximal Popliteal Arteries
Brief Title: ZENFlex-Registry to Evaluate the Outcome of Bare Metal Stent-assisted Angioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201805
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Atherosclerosis of Femoral Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZENFLEX stent Group (Experimental): subjects applying ZENFLEX peripheral stent system
  Interventions: Device: ZENFLEX peripheral stent system

INTERVENTIONS:
Device: ZENFLEX peripheral stent system — The ZENFLEX Peripheral Stent System is designed to deliver a self-expanding stent to the iliac artery, superficial femoral arteries and / or proximal popliteal arteries to improve luminal diameter. The self-expanding stent is composed of nickel titanium alloy (nitinol); contains a total of 12 tantalum / gold radiopaque markers and imparts an outward radial force on the luminal surface of the vessel to establish patency.

SUMMARY:
A prospective, multi-center, single-arm registry to evaluate the safety and efficacy of bare metal stent-assisted percutaneous transluminal angioplasty (PTA) in the treatment of superficial femoral and/or proximal popliteal artery (P1) lesions in patients with symptomatic peripheral artery disease

DETAILED DESCRIPTION:
The purpose of this registry is to collect acute and follow-up (up to 12 months) safety and efficacy data on the ZENFlex™ Peripheral Stent System in the stent-assisted angioplasty treatment of patients with de novo or restenotic lesion(s) of the native superficial femoral artery (SFA) and/or proximal popliteal artery (PPA, P1 segment) when used according to IFU. Up to 100 subjects will be enrolled in this study at up to 5 sites in Germany.

This study is a prospective, single-arm observational registry and does not include an active control arm. Therefore, no formal sample size calculation has been performed. All subjects will be evaluated at pre-discharge and during clinical follow-up visits 6 (182 ± 30 days) and 12 (365 ± 30 days) months post-procedure.

Primary endpoints are patency rate after one year and composite of freedom from device and procedure-related death through 12 months post procedure as well as freedom from both target limb major amputation and clinically-driven target lesion revascularization.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient is ≥ 18 years old at the time of consent. 2. Subject has provided written informed consent prior to participation in the study, understands the purpose of this study and agrees to comply with all protocol-specified examinations and follow-up appointments.

  3. Rutherford Classification Category 2-4. Subjects with Rutherford Class 2 have gone through a conservative therapy without success. 4. De novo stenotic, restenotic or occlusive lesion(s) located in the superficial femoral artery and/or proximal popliteal artery (P1 segment) suitable for stenting after PTA.

  5. Lesion location starts distal to CFA bifurcation (below origin of deep femoral artery) and should not extend beyond the P1 segment of the popliteal artery.

  6. Lesion(s) is/are located at least 2 cm from any stent if target limb was already previously stented.

  7. >70 % diameter stenosis or occlusion by visual angiographic estimate. 8. Patent inflow (treatment of inflow is allowed before treatment of the target lesion if successful).

  9. Patent ipsilateral popliteal artery (P2 and P3 segments) and at least 1 patent infrapopliteal artery in continuity to ankle. 10. Target reference vessel diameter ≥ 4 - ≤ 7.0 mm.

Exclusion Criteria:

* Patients will be excluded from the registry if any of the following criteria is met:

  1. Target Lesion previously tested with a stent or surgery.
  2. Rutherford Classification Category 0, 1, 5 or 6.
  3. Inability to tolerate antithrombotic or antiplatelet therapies.
  4. Known allergy or contraindication to contrast medium that, in the opinion of the investigator, can't be adequately pre-medicated.
  5. Non-dilatable severely calcified lesion.
  6. Known hypersensitivity to nitinol and/or its components (e.g. nickel, titanium).
  7. Acute or subacute thrombus in the target lesion.
  8. Documented life expectancy < 13 months
  9. Pregnancy or female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding.
  10. Other comorbidity risks which in the opinion of the investigator limit longevity or likelihood of compliance with protocol follow up.
  11. Myocardial infarction or stroke within 90 days prior to index procedure.
  12. Hypercoagulable state.
  13. Patient is currently enrolled in any other clinical investigational trial(s).
  14. Use of alternative therapy in target lesion during index procedure, e.g. atherectomy, lysis therapy, laser therapy, DES, re-entry-devices, cutting / scoring balloon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Patency rate | 12 (365 ± 30 days) months
  patency rate after one year defined as absence of clinically driven TLR (due to symptoms and drop of ABI of ≥ 20% or > 0.15 when compared to post-procedure baseline) or restenosis with PVR > 2.4 evaluated by Duplex Ultrasound
Procedure-related death | 12 (365 ± 30 days) months
  Composite of freedom from device and procedure-related death through 12 months post procedure as well as freedom from both target limb major amputation and clinically-driven target lesion revascularization。

SECONDARY OUTCOMES:
TLR rate at 6 and 12months | 6 (182 ± 30 days) and 12 (365 ± 30 days) months
  The ratio of either repeat percutaneous or surgical revascularization for target lesions
Sustained clinical improvement | 12 (365 ± 30 days) months
  an improvement shift in the Rutherford classification of one class in amputation and TVR free surviving patients at 12 months.
WIQ at 6 and 12 months | 6 (182 ± 30 days) and 12 (365 ± 30 days) months
  Walking capacity assessment by Walking Impairment Questionnaire (WIQ) at 6 and 12 months vs. baseline
Duplex-defined binary restenosis (PSVR >2.4) at 6 and 12 months or at any time of re-intervention | 6 (182 ± 30 days) and 12 (365 ± 30 days) months
  Duplex-defined binary restenosis (PSVR >2.4) of the target lesion post-procedure and at 6 and 12 months or at any time of re-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Study Director — Universitätsklinikum Leipzig; Annett Glanz, Principal Investigator — Diakoniekrankenhaus Halle
Locations (1):
- Popescu Diakoniekrankenhaus Halle gGmbH Klinik für Innere Medizin, Halle, Germany

IPD SHARING:
Plan to Share IPD: No